CLINICAL TRIAL: NCT04614623
Title: Defining the Role of Management Factors in Outcome Disparity in Pediatric T1D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Children's Hospital New Orleans, LA (Other)
Responsible Party: Principal Investigator, Stuart Chalew, Professor of Pediatrics, Director Pediatric Endocrine/Diabetes, Children's Hospital New Orleans, LA
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: R21DK118643 (NIH)
Record Dates: First submitted 2020-10-13; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Type1diabetes
Keywords: type1diabetes; health disparity; pediatrics; advanced hydbrid closed loop insulin pump; youth; HbA1c; teleconferencing; racial disparity; continuous glucose monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Current Diabetes Management Continued (No Intervention): Continued Insulin Delivery Method and Current Clinic Care of Diabetes
- Video Conferencing+Current Insulin Delivery (Experimental): Patients continue current insulin delivery modality but receive enhanced clinical management support via video conferencing link by diabetes coordinator
  Interventions: Other: Video conferencing Application
- AHCL pump without Video Conferencing (Experimental): Patients switch to use of an Advanced Hybrid Closed Loop pump without Video Conferencing standard support
  Interventions: Device: AHCL pump
- AHCL pump+Video Conferencing (Experimental): Patients will use Advanced Hybrid Closed Loop pump with enhanced clinical support via video conferencing
  Interventions: Device: AHCL pump; Other: Video conferencing Application

INTERVENTIONS:
Device: AHCL pump — Advanced Hybrid Closed Loop (AHCL) pump automatically adjusts insulin infusion rate of pump customized to patient's needs to reduce occurrence of hypo and hyperglycemia
  Arms: AHCL pump without Video Conferencing; AHCL pump+Video Conferencing
Other: Video conferencing Application — Video conferencing application will be used to enhance communication between participant and parent with the study certified diabetes educator (CDE) nurse coordinator. These individualized sessions will be designed to help the family with solving diabetes management problems to enhance glycemic control
  Arms: AHCL pump+Video Conferencing; Video Conferencing+Current Insulin Delivery

SUMMARY:
Type 1 diabetes (T1D), is associated with considerable risk of morbidity and mortality due to chronic hyperglycemia. Despite innovations in management, pediatric patients of African ancestry (AA) have been found to have persistently higher mean blood glucose (MBG) than European ancestry (EA) patients. The investigators hypothesize that an intervention using advanced insulin delivery technology together with home management will sustainably improve MBG to levels comparable to EA patients without increasing hypoglycemia.

The investigators will first perform a small "field trial" of the intervention in African American patients having T1D, with 8.5<HbA1c<12% aged 10-17 years. The primary intervention approach will use a combination of an advanced hybrid closed loop (AHCL) pump + enhanced home video management conferencing with study CDE nurse coordinator. Information gained in the "field trial" will be used to more specifically tailor the intervention in a randomized trial.

In the second part , the investigators will conduct a randomized trial of the study intervention in participants with the same clinical features as the field trial for a six month pilot period. Participants will be randomized into one of four groups. The special intervention group (AHCL+conferencing) group will be compared with a group using patient's current insulin management+followup, vs AHCL+without conferencing, vs patient's standard insulin management+conferencing. The investigators will compare HbA1c, MBG, time in glycemic range, ability to adhere with home management, satisfaction with management procedures between the groups.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D), one of the most prevalent incurable diseases of childhood, is associated with serious risk of morbidity and mortality due to the development of micro- and macrovascular complications. Complications can be prevented by treatment that achieves physiological or near physiological levels of glucose. Despite innovations in management over the past three decades, pediatric patients of African ancestry (AA) have had persistently higher HbA1c than patients of white, European ancestry (EA). Higher HbA1c in AA patients is associated with both higher acute and chronic morbidity and mortality compared to EA patients. Thus, racial disparity in glycemic outcome and the development of complications is a major unresolved challenge of current clinical pediatric diabetes treatment.

Multiple factors contribute to high-risk levels of mean blood glucose (MBG) in pediatric AA patients compared to EA. AA patients have less access to insulin pumps, perform glucose testing less often, have less contact with diabetes management staff, and may have difficulty relating to management staff due to cultural and socioeconomic differences. Greater occurrence of hypoglycemia is another obstacle to achieving optimal glucose control. These considerations have led us to hypothesize that an intervention targeting this group of major management obstacles will sustainably reduce MBG to levels comparable to EA patients without increased hypoglycemia. The investigators propose that an advanced hybrid closed loop (AHCL) pump system combined with frequent enhanced home video management conferencing (TECH) with the study CDE nurse coordinator will facilitate improvement of MBG and HbA1c, increase time in glycemic goal range, have minimal occurrence of hypoglycemia, and improve patient satisfaction with management.

Part 1: The investigators will first pre-test the intervention approach in ten participants using a combination of an advanced hybrid closed loop (AHCL) pump system + home video conferences with the study CDE nurse coordinator to enhance home management. Basic inclusion criterion will be self-identification as African American ethnicity, having T1D, 8.5<HbA1c<12%, age 10-17 years. The field trial will be for a 4 week period. THe investigators will use feedback and experience during the "field trial" from patients, parents and the study coordinator to refine the intervention and reduce patient problems with the technology, enhance its effectiveness improve participant adherence to management. This information will help guide/refine the design and use of the technologies in a randomized intervention trial (Part 2). Participants may choose to continue using the technologies after the initial 4 week Field Trial period for up to 6 months. AHCL must be returned at the end of participation.

Part 2: The investigators will conduct a randomized intervention trial in a factorial four group design comparing outcome measures in participants assigned to the combined AHCL+conferencing, versus use of AHCL or conferencing alone versus usual care. Basic inclusion criterion will be self-identification as African American ethnicity, having T1D, 8.5<HbA1c<12%, age 10-17 years. Outcome measures will be assessed at 3 and 6 month study visits. The major outcome metric will be HbA1c. In addition mean blood glucose (MBG), time in range, frequency of hyper/hypoglycemia, quality of life and treatment satisfaction will be compared between groups, Participation will be concluded at the 6 month visit. AHCL must be returned at the end of participation.

ELIGIBILITY:
Inclusion Criteria:

* T1D as defined by:

  * Typical clinical presentation at diagnosis
  * Prior documentation of one or more anti-pancreatic antibodies
  * Requiring >0.3 units/kg/d insulin therapy
  * On no oral hypoglycemic agents concurrently
  * Body mass index (BMI) <90% for age and gender
* T1D duration of ≥ 6 months
* Self-identification as of African ancestry (AA)
* Age 10-17 years inclusive
* Pre-recruitment HbA1c 8.6-12%
* Glucose meter MBG ≥ 200 mg/dL
* Have smartphone/tablet/computer for conferencing
* Willingness to download and use the app for conferencing
* Willingness to be randomized to one of the clinical arms of the study (for Randomized intervention trial)
* Willingness and ability to wear pump and sensor, maintain equipment, and upload data from the system
* In stable living environment with a parent or guardian trained and able to recognize and intervene in diabetes emergency such as DKA or hypoglycemia
* Willingness to attend clinic visits during study at 3 and 6 month intervals

Exclusion Criteria:

* Unwillingness or inability to be randomized and/or participate in study procedures
* Pregnancy/plans to become pregnant/immediate post pregnancy and breast feeding
* Smoking, alcohol use, illicit drug use
* Severe psychiatric illness of patient or parent/guardian
* More than one (1) episode of diabetic ketoacidosis (DKA) in the past year
* Inability to wear sensor and/or pump catheter
* Known allergy to medical adhesives
* Less than two (2) clinic visits in the past year
* Absence of anti-pancreatic antibodies at diagnosis
* BMI ≥90%
* Hypoglycemic unawareness associated with severe episodes of hypoglycemia
* Insulin requirement <0.3 units/kg/d
* On hypoglycemic agent besides insulin within prior 6 months or other medication which in the judgment of the investigator may be a contraindication to participation in the study.
* Other chronic illness or condition besides diabetes (exception for hypothyroidism if stable on thyroxine replacement therapy) that would interfere in patient or family's participation in the study, or would influence metabolic control or HbA1c interpretation
* Inability to participate in "run-in" pre-randomization activities for randomized trial

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) Change From Baseline to 6 months (End of study) | Change in HbA1c will be assessed from baseline to the HbA1c at 6 months (end of study)
  Hemoglobin A1c (Glycated hemoglobin)

SECONDARY OUTCOMES:
Mean blood glucose (MBG) Change From Baseline to 6 months (End of study) | Change in MBG will be assessed at baseline and compared with 6 month measure (study end)
  Mean glucose levels as estimated from recorded glucose meter and sensor data

OTHER OUTCOMES:
Time in Glucose Range Change From Baseline to 6 months (End of study) | Cnge in Percent of Time in and out of glucose range at Baseline will be compared with 6 month measurement (study end)
  Percent Time Spent in Hyper/Hypo and Goal glucose ranges during the study
DSMP-SR Change from Baseline to 6 months (End of Study) | Assessment of Change: Baseline will be compared with 6 month measure (study end)
  Diabetes Self-Management Profile
PedsQL-Diabetes Module Change from Baseline to 6 months (study end) | Assessment of Change: Baseline compared with 6 month measure (study end)
  Pediatric Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Chalew, M.D., Principal Investigator — Children's Hospital of New Orleans/ LSUHSC Dept of Pediatrics
Locations (1):
- Children's Hospital of New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naranjo D, Schwartz DD, Delamater AM. Diabetes in ethnically diverse youth: disparate burden and intervention approaches. Curr Diabetes Rev. 2015;11(4):251-60. doi: 10.2174/1573399811666150421115846. PMID 25901501
- [Background] Bergenstal RM, Garg S, Weinzimer SA, Buckingham BA, Bode BW, Tamborlane WV, Kaufman FR. Safety of a Hybrid Closed-Loop Insulin Delivery System in Patients With Type 1 Diabetes. JAMA. 2016 Oct 4;316(13):1407-1408. doi: 10.1001/jama.2016.11708. No abstract available. PMID 27629148
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Service FJ, O'Brien PC. The relation of glycaemia to the risk of development and progression of retinopathy in the Diabetic Control and Complications Trial. Diabetologia. 2001 Oct;44(10):1215-20. doi: 10.1007/s001250100635. PMID 11692169
- [Background] Ryan CM, van Duinkerken E, Rosano C. Neurocognitive consequences of diabetes. Am Psychol. 2016 Oct;71(7):563-576. doi: 10.1037/a0040455. PMID 27690485
- [Background] Rewers MJ, Pillay K, de Beaufort C, Craig ME, Hanas R, Acerini CL, Maahs DM; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Assessment and monitoring of glycemic control in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:102-14. doi: 10.1111/pedi.12190. No abstract available. PMID 25182311
- [Background] American Diabetes Association. Standards of medical care in diabetes: children and adolescents. Diabetes Care. 2015;38 (Supplement 1):S70-S6.
- [Background] Hanson CL, Henggeler SW, Burghen GA. Race and sex differences in metabolic control of adolescents with IDDM: a function of psychosocial variables? Diabetes Care. 1987 May-Jun;10(3):313-8. doi: 10.2337/diacare.10.3.313. PMID 3595397
- [Background] Auslander WF, Anderson BJ, Bubb J, Jung KC, Santiago JV. Risk factors to health in diabetic children: a prospective study from diagnosis. Health Soc Work. 1990 May;15(2):133-42. doi: 10.1093/hsw/15.2.133. PMID 2365239
- [Background] Delamater AM, Albrecht DR, Postellon DC, Gutai JP. Racial differences in metabolic control of children and adolescents with type I diabetes mellitus. Diabetes Care. 1991 Jan;14(1):20-5. doi: 10.2337/diacare.14.1.20. PMID 1991431
- [Background] Chalew SA, Gomez R, Butler A, Hempe J, Compton T, Mercante D, Rao J, Vargas A. Predictors of glycemic control in children with type 1 diabetes: the importance of race. J Diabetes Complications. 2000 Mar-Apr;14(2):71-7. doi: 10.1016/s1056-8727(00)00072-6. PMID 10959068
- [Background] Petitti DB, Klingensmith GJ, Bell RA, Andrews JS, Dabelea D, Imperatore G, Marcovina S, Pihoker C, Standiford D, Waitzfelder B, Mayer-Davis E; SEARCH for Diabetes in Youth Study Group. Glycemic control in youth with diabetes: the SEARCH for diabetes in Youth Study. J Pediatr. 2009 Nov;155(5):668-72.e1-3. doi: 10.1016/j.jpeds.2009.05.025. Epub 2009 Jul 29. PMID 19643434
- [Background] Kamps JL, Hempe JM, Chalew SA. Racial disparity in A1C independent of mean blood glucose in children with type 1 diabetes. Diabetes Care. 2010 May;33(5):1025-7. doi: 10.2337/dc09-1440. Epub 2010 Feb 25. PMID 20185743
- [Background] Redondo MJ, Connor CG, Ruedy KJ, Beck RW, Kollman C, Wood JR, Buckingham B, Klingensmith GJ, Silverstein J, Tamborlane WV; Pediatric Diabetes Consortium. Pediatric Diabetes Consortium Type 1 Diabetes New Onset (NeOn) Study: factors associated with HbA1c levels one year after diagnosis. Pediatr Diabetes. 2014 Jun;15(4):294-302. doi: 10.1111/pedi.12061. Epub 2013 Jul 24. PMID 23889707
- [Background] Willi SM, Miller KM, DiMeglio LA, Klingensmith GJ, Simmons JH, Tamborlane WV, Nadeau KJ, Kittelsrud JM, Huckfeldt P, Beck RW, Lipman TH; T1D Exchange Clinic Network. Racial-ethnic disparities in management and outcomes among children with type 1 diabetes. Pediatrics. 2015 Mar;135(3):424-34. doi: 10.1542/peds.2014-1774. PMID 25687140
- [Background] Dabelea D, Rewers A, Stafford JM, Standiford DA, Lawrence JM, Saydah S, Imperatore G, D'Agostino RB Jr, Mayer-Davis EJ, Pihoker C; SEARCH for Diabetes in Youth Study Group. Trends in the prevalence of ketoacidosis at diabetes diagnosis: the SEARCH for diabetes in youth study. Pediatrics. 2014 Apr;133(4):e938-45. doi: 10.1542/peds.2013-2795. Epub 2014 Mar 31. PMID 24685959
- [Background] Saydah S, Imperatore G, Cheng Y, Geiss LS, Albright A. Disparities in Diabetes Deaths Among Children and Adolescents - United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2017 May 19;66(19):502-505. doi: 10.15585/mmwr.mm6619a4. PMID 28520705
- [Background] Secrest AM, Becker DJ, Kelsey SF, LaPorte RE, Orchard TJ. All-cause mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes: the Allegheny County type 1 diabetes registry. Diabetes Care. 2010 Dec;33(12):2573-9. doi: 10.2337/dc10-1170. PMID 21115767
- [Background] US Department of Health and Human Services. Initiative to eliminate racial disparities in health. 2003.
- [Background] Paris CA, Imperatore G, Klingensmith G, Petitti D, Rodriguez B, Anderson AM, Schwartz ID, Standiford DA, Pihoker C. Predictors of insulin regimens and impact on outcomes in youth with type 1 diabetes: the SEARCH for Diabetes in Youth study. J Pediatr. 2009 Aug;155(2):183-9.e1. doi: 10.1016/j.jpeds.2009.01.063. Epub 2009 Apr 24. PMID 19394043
- [Background] Lin MH, Connor CG, Ruedy KJ, Beck RW, Kollman C, Buckingham B, Redondo MJ, Schatz D, Haro H, Lee JM, Tamborlane WV, Wood JR; Pediatric Diabetes Consortium. Race, socioeconomic status, and treatment center are associated with insulin pump therapy in youth in the first year following diagnosis of type 1 diabetes. Diabetes Technol Ther. 2013 Nov;15(11):929-34. doi: 10.1089/dia.2013.0132. Epub 2013 Jul 19. PMID 23869706
- [Background] Coulon SJ, Velasco-Gonzalez C, Scribner R, Park CL, Gomez R, Vargas A, Stender S, Zabaleta J, Clesi P, Chalew SA, Hempe JM. Racial differences in neighborhood disadvantage, inflammation and metabolic control in black and white pediatric type 1 diabetes patients. Pediatr Diabetes. 2017 Mar;18(2):120-127. doi: 10.1111/pedi.12361. Epub 2016 Jan 18. PMID 26783014
- [Background] Auslander WF, Thompson S, Dreitzer D, White NH, Santiago JV. Disparity in glycemic control and adherence between African-American and Caucasian youths with diabetes. Family and community contexts. Diabetes Care. 1997 Oct;20(10):1569-75. doi: 10.2337/diacare.20.10.1569. PMID 9314637
- [Background] Chalew S, Gomez R, Vargas A, Kamps J, Jurgen B, Scribner R, Hempe J. Hemoglobin A1c, frequency of glucose testing and social disadvantage: Metrics of racial health disparity in youth with type 1 diabetes. J Diabetes Complications. 2018 Dec;32(12):1085-1090. doi: 10.1016/j.jdiacomp.2018.02.008. Epub 2018 Aug 10. PMID 30318164
- [Background] Chalew SA, Harrison J, Berry S. Achievement of glycemic outcome goals in pediatric diabetes: the impact of staff number. J La State Med Soc. 2008 Nov-Dec;160(6):328-32. PMID 19283981
- [Background] Valenzuela JM, Seid M, Waitzfelder B, Anderson AM, Beavers DP, Dabelea DM, Dolan LM, Imperatore G, Marcovina S, Reynolds K, Yi-Frazier J, Mayer-Davis EJ; SEARCH for Diabetes in Youth Study Group. Prevalence of and disparities in barriers to care experienced by youth with type 1 diabetes. J Pediatr. 2014 Jun;164(6):1369-75.e1. doi: 10.1016/j.jpeds.2014.01.035. Epub 2014 Feb 25. PMID 24582008
- [Background] Valenzuela JM, Smith LB, Stafford JM, D'Agostino RB Jr, Lawrence JM, Yi-Frazier JP, Seid M, Dolan LM. Shared decision-making among caregivers and health care providers of youth with type 1 diabetes. J Clin Psychol Med Settings. 2014 Sep;21(3):234-43. doi: 10.1007/s10880-014-9400-9. PMID 24952739
- [Background] Lipman TH, Murphy KM, Kumanyika SK, Ratcliffe SJ, Jawad AF, Ginsburg KR. Racial differences in parents' perceptions of factors important for children to live well with diabetes. Diabetes Educ. 2012 Jan-Feb;38(1):58-66. doi: 10.1177/0145721711427454. Epub 2011 Dec 6. PMID 22146789
- [Background] Hamdan MA, Hempe JM, Velasco-Gonzalez C, Gomez R, Vargas A, Chalew S. Differences in Red Blood Cell Indices Do Not Explain Racial Disparity in Hemoglobin A1c in Children with Type 1 Diabetes. J Pediatr. 2016 Sep;176:197-9. doi: 10.1016/j.jpeds.2016.03.068. Epub 2016 May 4. PMID 27156184
- [Background] Bergenstal RM, Gal RL, Connor CG, Gubitosi-Klug R, Kruger D, Olson BA, Willi SM, Aleppo G, Weinstock RS, Wood J, Rickels M, DiMeglio LA, Bethin KE, Marcovina S, Tassopoulos A, Lee S, Massaro E, Bzdick S, Ichihara B, Markmann E, McGuigan P, Woerner S, Ecker M, Beck RW; T1D Exchange Racial Differences Study Group. Racial Differences in the Relationship of Glucose Concentrations and Hemoglobin A1c Levels. Ann Intern Med. 2017 Jul 18;167(2):95-102. doi: 10.7326/M16-2596. Epub 2017 Jun 13. PMID 28605777
- [Background] Chalew S, Hamdan M. Racial disparity in HbA1c persists when fructosamine is used as a surrogate for mean blood glucose in youth with type 1 diabetes. Pediatr Diabetes. 2018 Nov;19(7):1243-1248. doi: 10.1111/pedi.12696. Epub 2018 Aug 21. PMID 29808574
- [Background] Chalew SA. The continuing challenge of outcome disparities in children with diabetes. Pediatrics. 2015 Mar;135(3):552-3. doi: 10.1542/peds.2014-4136. No abstract available. PMID 25687141
- [Background] Redondo MJ, Libman I, Cheng P, Kollman C, Tosur M, Gal RL, Bacha F, Klingensmith GJ, Clements M; Pediatric Diabetes Consortium. Racial/Ethnic Minority Youth With Recent-Onset Type 1 Diabetes Have Poor Prognostic Factors. Diabetes Care. 2018 May;41(5):1017-1024. doi: 10.2337/dc17-2335. Epub 2018 Mar 1. PMID 29496742
- [Background] Wild D, von Maltzahn R, Brohan E, Christensen T, Clauson P, Gonder-Frederick L. A critical review of the literature on fear of hypoglycemia in diabetes: Implications for diabetes management and patient education. Patient Educ Couns. 2007 Sep;68(1):10-5. doi: 10.1016/j.pec.2007.05.003. Epub 2007 Jun 19. PMID 17582726
- [Background] Dabelea D, Mayer-Davis EJ, Saydah S, Imperatore G, Linder B, Divers J, Bell R, Badaru A, Talton JW, Crume T, Liese AD, Merchant AT, Lawrence JM, Reynolds K, Dolan L, Liu LL, Hamman RF; SEARCH for Diabetes in Youth Study. Prevalence of type 1 and type 2 diabetes among children and adolescents from 2001 to 2009. JAMA. 2014 May 7;311(17):1778-86. doi: 10.1001/jama.2014.3201. PMID 24794371
- [Background] Mayer-Davis EJ, Lawrence JM, Dabelea D, Divers J, Isom S, Dolan L, Imperatore G, Linder B, Marcovina S, Pettitt DJ, Pihoker C, Saydah S, Wagenknecht L; SEARCH for Diabetes in Youth Study. Incidence Trends of Type 1 and Type 2 Diabetes among Youths, 2002-2012. N Engl J Med. 2017 Apr 13;376(15):1419-1429. doi: 10.1056/NEJMoa1610187. PMID 28402773
- [Background] Fairchild JM, Hing SJ, Donaghue KC, Bonney MA, Fung AT, Stephens MM, Mitchell P, Howard NJ, Silink M. Prevalence and risk factors for retinopathy in adolescents with type 1 diabetes. Med J Aust. 1994 Jun 20;160(12):757-62. doi: 10.5694/j.1326-5377.1994.tb125943.x. PMID 8208191
- [Background] Donaghue KC, Fairchild JM, Craig ME, Chan AK, Hing S, Cutler LR, Howard NJ, Silink M. Do all prepubertal years of diabetes duration contribute equally to diabetes complications? Diabetes Care. 2003 Apr;26(4):1224-9. doi: 10.2337/diacare.26.4.1224. PMID 12663601
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Research Group; Nathan DM, Zinman B, Cleary PA, Backlund JY, Genuth S, Miller R, Orchard TJ. Modern-day clinical course of type 1 diabetes mellitus after 30 years' duration: the diabetes control and complications trial/epidemiology of diabetes interventions and complications and Pittsburgh epidemiology of diabetes complications experience (1983-2005). Arch Intern Med. 2009 Jul 27;169(14):1307-16. doi: 10.1001/archinternmed.2009.193. PMID 19636033
- [Background] Molitch ME, Steffes M, Sun W, Rutledge B, Cleary P, de Boer IH, Zinman B, Lachin J; Epidemiology of Diabetes Interventions and Complications Study Group. Development and progression of renal insufficiency with and without albuminuria in adults with type 1 diabetes in the diabetes control and complications trial and the epidemiology of diabetes interventions and complications study. Diabetes Care. 2010 Jul;33(7):1536-43. doi: 10.2337/dc09-1098. Epub 2010 Apr 22. PMID 20413518
- [Background] Polak JF, Backlund JY, Cleary PA, Harrington AP, O'Leary DH, Lachin JM, Nathan DM; DCCT/EDIC Research Group. Progression of carotid artery intima-media thickness during 12 years in the Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) study. Diabetes. 2011 Feb;60(2):607-13. doi: 10.2337/db10-0296. PMID 21270271
- [Background] Khanolkar AR, Amin R, Taylor-Robinson D, Viner RM, Warner JT, Stephenson T. Young people with Type 1 diabetes of non-white ethnicity and lower socio-economic status have poorer glycaemic control in England and Wales. Diabet Med. 2016 Nov;33(11):1508-1515. doi: 10.1111/dme.13079. Epub 2016 Feb 23. PMID 26802317
- [Background] Tull ES, Barinas E. A twofold excess mortality among black compared with white IDDM patients in Allegheny county, Pennsylvania. Pittsburgh DERI Mortality Study Group. Diabetes Care. 1996 Dec;19(12):1344-7. doi: 10.2337/diacare.19.12.1344. PMID 8941461
- [Background] Secrest AM, Becker DJ, Kelsey SF, Laporte RE, Orchard TJ. Cause-specific mortality trends in a large population-based cohort with long-standing childhood-onset type 1 diabetes. Diabetes. 2010 Dec;59(12):3216-22. doi: 10.2337/db10-0862. Epub 2010 Aug 25. PMID 20739685
- [Background] Dias RP, Brown F, Wyatt C, Cheema S, Allgrove J, Amin R. The effect of insulin intensification in children and young persons with Type 1 diabetes differs in relation to ethnic group; a prospective observational study. Diabet Med. 2013 Apr;30(4):495-501. doi: 10.1111/dme.12022. PMID 22998464
- [Background] Markowitz JT, Volkening LK, Laffel LM. Care utilization in a pediatric diabetes clinic: cancellations, parental attendance, and mental health appointments. J Pediatr. 2014 Jun;164(6):1384-9. doi: 10.1016/j.jpeds.2014.01.045. Epub 2014 Mar 6. PMID 24612905
- [Background] Messer LH, Forlenza GP, Sherr JL, Wadwa RP, Buckingham BA, Weinzimer SA, Maahs DM, Slover RH. Optimizing Hybrid Closed-Loop Therapy in Adolescents and Emerging Adults Using the MiniMed 670G System. Diabetes Care. 2018 Apr;41(4):789-796. doi: 10.2337/dc17-1682. Epub 2018 Feb 14. PMID 29444895
- [Background] Rustad JK, Musselman DL, Skyler JS, Matheson D, Delamater A, Kenyon NS, Caceda R, Nemeroff CB. Decision-making in diabetes mellitus type 1. J Neuropsychiatry Clin Neurosci. 2013 Winter;25(1):40-50. doi: 10.1176/appi.neuropsych.12010016. PMID 23487192
- [Background] Hilliard ME, Rohan JM, Rausch JR, Delamater A, Pendley JS, Drotar D. Patterns and predictors of paternal involvement in early adolescents' type 1 diabetes management over 3 years. J Pediatr Psychol. 2014 Jan-Feb;39(1):74-83. doi: 10.1093/jpepsy/jst067. Epub 2013 Sep 6. PMID 24013966
- [Background] Lord JH, Young MT, Gruhn MA, Grey M, Delamater AM, Jaser SS. Effect of race and marital status on mothers' observed parenting and adolescent adjustment in youth with type 1 diabetes. J Pediatr Psychol. 2015 Jan-Feb;40(1):132-43. doi: 10.1093/jpepsy/jsu078. Epub 2014 Sep 23. PMID 25248850
- [Background] Messer LH, Forlenza GP, Wadwa RP, Weinzimer SA, Sherr JL, Hood KK, Buckingham BA, Slover RH, Maahs DM. The dawn of automated insulin delivery: A new clinical framework to conceptualize insulin administration. Pediatr Diabetes. 2018 Feb;19(1):14-17. doi: 10.1111/pedi.12535. Epub 2017 Jun 27. No abstract available. PMID 28656656
- [Background] Sherr JL, Cengiz E, Palerm CC, Clark B, Kurtz N, Roy A, Carria L, Cantwell M, Tamborlane WV, Weinzimer SA. Reduced hypoglycemia and increased time in target using closed-loop insulin delivery during nights with or without antecedent afternoon exercise in type 1 diabetes. Diabetes Care. 2013 Oct;36(10):2909-14. doi: 10.2337/dc13-0010. Epub 2013 Jun 11. PMID 23757427
- [Background] Rodbard D. Continuous Glucose Monitoring: A Review of Recent Studies Demonstrating Improved Glycemic Outcomes. Diabetes Technol Ther. 2017 Jun;19(S3):S25-S37. doi: 10.1089/dia.2017.0035. PMID 28585879
- [Background] Dougherty JP, Lipman TH, Hyams S, Montgomery KA. Telemedicine for adolescents with type 1 diabetes. West J Nurs Res. 2014 Oct;36(9):1199-221. doi: 10.1177/0193945914528387. Epub 2014 Apr 1. PMID 24695401
- [Background] Davis RM, Hitch AD, Salaam MM, Herman WH, Zimmer-Galler IE, Mayer-Davis EJ. TeleHealth improves diabetes self-management in an underserved community: diabetes TeleCare. Diabetes Care. 2010 Aug;33(8):1712-7. doi: 10.2337/dc09-1919. Epub 2010 May 18. PMID 20484125
- [Background] Wood CL, Clements SA, McFann K, Slover R, Thomas JF, Wadwa RP. Use of Telemedicine to Improve Adherence to American Diabetes Association Standards in Pediatric Type 1 Diabetes. Diabetes Technol Ther. 2016 Jan;18(1):7-14. doi: 10.1089/dia.2015.0123. Epub 2015 Aug 21. PMID 26295939
- [Background] Resnicow K, Baranowski T, Ahluwalia JS, Braithwaite RL. Cultural sensitivity in public health: defined and demystified. Ethn Dis. 1999 Winter;9(1):10-21. PMID 10355471
- [Background] Wysocki T, Buckloh LM, Antal H, Lochrie A, Taylor A. Validation of a self-report version of the diabetes self-management profile. Pediatr Diabetes. 2012 Aug;13(5):438-43. doi: 10.1111/j.1399-5448.2011.00823.x. Epub 2011 Oct 3. PMID 21967680
- [Background] Laffel LM, Connell A, Vangsness L, Goebel-Fabbri A, Mansfield A, Anderson BJ. General quality of life in youth with type 1 diabetes: relationship to patient management and diabetes-specific family conflict. Diabetes Care. 2003 Nov;26(11):3067-73. doi: 10.2337/diacare.26.11.3067. PMID 14578241
- [Background] Varni JW, Burwinkle TM, Jacobs JR, Gottschalk M, Kaufman F, Jones KL. The PedsQL in type 1 and type 2 diabetes: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales and type 1 Diabetes Module. Diabetes Care. 2003 Mar;26(3):631-7. doi: 10.2337/diacare.26.3.631. PMID 12610013